CLINICAL TRIAL: NCT07181616
Title: Feasibility, Acceptability, and Preliminary Efficacy of an HIV Prevention Intervention for Older Black Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laneshia Conner (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Laneshia Conner, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 78084; K01AG092253-01A1 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Health Risk Behaviors
Keywords: HIV; Health Education; Health Equity
MeSH Terms: conditions — Health Risk Behaviors; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapted W2W (Experimental): HIV intervention focused on aging-related HIV knowledge, identifying HIV prevention practices, and reducing HIV transmission. Intervention given in four, 2 hour educational sessions with a fifth booster session and a final follow up session.
  Interventions: Behavioral: Adapted W2W
- Waitlist Control (Active Comparator): This group will receive the intervention 8 weeks after the W2W intervention group completes their follow-up and in the same pattern.
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Adapted W2W — HIV education sessions and questionnaires.
  Arms: Adapted W2W
Behavioral: Waitlist Control — HIV education sessions and questionnaires given 4 weeks after W2W intervention.
  Arms: Waitlist Control

SUMMARY:
The goal of this clinical trial is to learn whether a group-based HIV prevention program can improve HIV knowledge, prevention behaviors, and testing in older Black women aged 50 and older who live in subsidized housing. The study focuses on improving how HIV prevention programs address the unique needs and life experiences of older Black women.

The main questions it aims to answer are:

Can a revised HIV prevention intervention tailored to reproductive health histories improve HIV knowledge, condom use, and testing in older Black women?

Is the intervention feasible, acceptable, and engaging for participants?

The PI will compare a group of participants receiving the Woman-2-Woman (W2W) intervention to a wait-listed control group to see if the intervention leads to better HIV prevention outcomes.

Participants will:

Join a group-based HIV prevention program designed for older Black women

Be randomly assigned to either:

Start the intervention right away, or

Join a waitlist and start the program 4 weeks later

Take part in four weekly sessions that include group discussions, education, and skill-building activities

Share information about their reproductive health histories and sexual health decisions during focus groups or surveys

Complete questionnaires at the start, after the program ends, and 4 weeks later to assess HIV knowledge, condom use, and testing behavior

This research aims to create a culturally tailored, evidence-based HIV intervention that fits the lives and needs of older Black women and can be used in future, larger studies.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age
* A resident of Selected sites
* A MOCA score of less than 24
* Self-identifying as an African American woman
* English speaking

Exclusion Criteria:

* Pre-menopausal
* Cognitive impairment

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Feasibility will be measured by recruitment rate (number of participants who sign the informed consent divided by those participants who meet the eligibility criteria)
Acceptability | Assessed at weeks 1,2,3,4, 8 and 12
  Acceptability will be measured by program satisfaction evaluations. Participants rate statements (1-5) with higher scores equating to greater satisfaction.
Retention Rate | Baseline (week 1) and Post-Intervention (Week 8)
  Feasibility will also be measured by retention rate (number of participants who complete all 4 sessions divided by those participants who signed the informed consent)
Change in HIV Knowledge | Baseline (week 1), Post-Intervention (Week 8), and Study completion (Week 12)
  HIV knowledge will be measured by the HIV-KQ-18. Scores range from 0-18 with higher scores equating to greater HIV knowledge.
Change in Condom-use self-efficacy (CUSES) | Baseline (week 1), Post-Intervention (Week 8), and Study completion (Week 12)
  CUSES is a 28 item scale that will assess behavioral intentions and past behavior related to feelings about purchasing, using, and negotiating use of condoms with a new partner. Each item has a 5-point response format ranging from 0 (strongly disagree) to 4 (strongly agree). After reversing negatively worded items, scores range from 0-112 (with higher scores indicating more self-efficacy).
Change in H-AGE scale | Baseline (week 1), Post-Intervention (Week 8), and Study completion (Week 12)
  The H-AGE scale is a gender and aging specific HIV knowledge scale with 6 items that assess participants knowledge of gender and age related issues regarding HIV. Q1 is a true/false question; Q2 & 3 are multiple choice questions; Q4 is rating of strongly disagree (1) to strongly agree (5); Q5 is rating very comfortable (1)to very uncomfortable (5); Q6 they select one from the following (positive, negative, mixed, neutral)

CONTACTS AND LOCATIONS:
Overall Officials: Laneshia Conner, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No